CLINICAL TRIAL: NCT01158326
Title: Evaluation of Efficacy and Safety of Oral Solution Paracetamol, Maleate Chlorpheniramine and Phenylephrine Hydrochloride in Reducing Symptoms of Common Cold and Flu: a Double-blind
Brief Title: Evaluation of Efficacy and Safety of Oral Solution Resfenol in Reducing Symptoms of Common Cold And Flu
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: PROFESSOR DOUTOR PAULO DORNELLES PICON, HOSPITAL DE CLINICAS DE PORTO ALEGRE
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-542
Record Dates: First submitted 2010-02-25; First posted 2010-07-08 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Common Cold; Influenza
Keywords: reducing symptoms; events; Common Cold; flu syndrome; Symptomatic treatment of the Common Cold and Flu syndrome
MeSH Terms: conditions — Common Cold; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resfenol Solution oral (Active Comparator): Acetaminophen, chlorpheniramine maleate, phenylephrine hydrochloride active drug
  Interventions: Drug: Resfenol
- Placebo (Placebo Comparator): Placebo oral solution
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Resfenol — Paracetamol (acetaminophen), chlorpheniramine maleate, phenylephrine hydrochloride.
  10 ml of oral solution acetaminophen, chlorpheniramine maleate, phenylephrine hydrochloride every 6 hours for 48 hours.
  Other Names: Antigripal
  Arms: Resfenol Solution oral
Other: Placebo — 10 ml of oral placebo every 6 hours for 48 hours
  Other Names: Placebo Antigripal
  Arms: Placebo

SUMMARY:
This study aimed to evaluate the efficacy and safety of the oral solution of paracetamol, chlorpheniramine maleate and phenylephrine hydrochloride in reducing symptoms of flu and the common cold. There will be a randomized, double-blind, placebo-controlled trial. Will be included 216 subjects, male or female, aged greater than 12 and less than or equal to 60 years, irrespective of color and / or race with symptoms of recent onset, for more than 6 hours and less than 48 hours length, characterizing Common Cold and / or Influenza.

After clinical evaluation and laboratory research subjects will be randomized to receive active drug or placebo, 10 ml oral solution every 6 hours for 48 hours. The follow-up visits will be held on 2 (24 hours after first intervention) and in 3 days (48 hours after first intervention).

The outcomes to assess the effectiveness so far consist of the scores of symptoms and to assess the safety of the drug will be accompanied by the emergence of adverse events.

DETAILED DESCRIPTION:
Infections of upper respiratory tract are common in the population, and its treatment, in most cases involves the use of symptomatic drugs. Paracetamol is used as an analgesic and antipyretic, while chlorpheniramine is an antihistamine and a vasoconstrictor phenylephrine decongestant function. This study aimed to evaluate the efficacy and safety of the oral solution of paracetamol, chlorpheniramine maleate and phenylephrine hydrochloride in reducing symptoms of flu and the common cold. There will be a randomized, double-blind, placebo-controlled trial. Volunteers will be recruited through posters down at the Hospital de Clinicals de Porto Alegre, and care in the public hospital network, which will undergo a screening questionnaire on first contact. With a statistical power of 80% and the possibility of random error of 5% should be followed in this study 194 subjects. Whereas a loss of up to 10% will be included 216 subjects, male or female, aged greater than 12 and less than or equal to 60 years, irrespective of color and / or race with symptoms of recent onset, for more than 6 hours and less than 48 hours, characterizing one of the following conditions: Common Cold, which consists of at least 3 symptoms among the 10 following: sneezing, rhinorrhea, nasal congestion, headache, muscle pain, throat discomfort, pain throat, dysphonia, cough, fever, and these moderate or severe using a scale of severity of symptoms of 4 points (0 = none, 1 = mild, 2 = moderate, 3 = severe) and / or Influenza consisting fever of at least 38.1 ° C and headache of moderate or severe or myalgia / arthralgia moderate or severe using a scale of severity of symptoms of 4 points (0 = none, 1 = mild, 2 = moderate , 3 = severe). Will be included only subjects who agree with the Terms of Consent. Not be included in the study pregnant women or infants with known hypersensitivity to components of the formula, or research subjects that are experiencing chronic active or exacerbated. After clinical evaluation and laboratory research subjects will be randomized to receive active drug or placebo, 10 ml oral solution every 6 hours for 48 hours. Be provided paracetamol rescue co-intervention. Study subjects will receive a diary containing questionnaires of symptoms. The follow-up visits will be held on 2 (24 hours after first intervention) and in 3 days (48 hours after first intervention). The outcomes to assess the effectiveness so far consist of scores of symptoms, rescue medication use, improvement of fever, subjective evaluation of palatability and tolerance and treatment compliance. To evaluate the safety of the drug will be accompanied by the emergence of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Men or women older than 12 years and less than or equal to 60 years, without distinction of color and / or race.
* Presenting symptoms of recent onset, for more than 6 hours and less than 48 hours, characterizing one of the following conditions:

Common cold, which consists of at least 3 symptoms among the 10 following: sneezing, rhinorrhea, nasal congestion, headache, muscle pain, discomfort in the throat, sore throat, dysphonia, cough, fever, and these moderate or severe by a scale of severity of symptoms of 4 points (0 = none, 1 = mild, 2 = moderate, 3 = severe),

OR

Flu-like symptoms consisting of fever of at least 38.1 ° C and headache of moderate or severe or myalgia / arthralgia moderate or severe using a scale of severity of symptoms of 4 points (0 = none, 1 = mild, 2 = moderate, 3 = severe).

* Adequate contraception, a woman of childbearing age.
* Do not use any other drugs for the treatment of clinical symptoms, except in cases of urgency, and immediate notification to the investigator. Patients with chronic diseases being treated with monotherapy, stable over the last three months, may be included after medical evaluation.
* Good ability of understanding and cooperation.
* Agreement with the informed consent consent (IC).
* Assessment exams, the medical criteria:

  * Pregnancy test (rapid urine), a woman of childbearing age, performed prior to inclusion;
  * 12-lead electrocardiogram performed during the consultation
  * Complete blood count and platelet count, serum creatinine, serum urea, serum sodium, serum potassium, total bilirubin and fractions, gamma-glutamyltransferase, alkaline phosphatase, aspartate aminotransferase (AST), alanine aminotransferase (ALT), prothrombin time , amylase, blood glucose (if possible in eight hours of fasting), TSH, urinalysis I, chorionic gonadotropin (β-HCG)

Exclusion Criteria:

* Pregnant or lactating women
* Known hypersensitivity to components of the formula of the drug solution active
* Use of alcohol or illicit drug use
* Use of monoamine oxidase (MAO) or barbiturates
* Diagnosis of allergic rhinitis or perennial activity
* Presenting the diagnosis of any disease or active acute exacerbated chronic disease (not compensated), including hypertension, ischemic heart disease, narrow-angle glaucoma, symptomatic prostatic hyperplasia, chronic renal failure, liver diseases, infectious tracheobronchitis presumably bacterial pneumonia, streptococcal pharyngitis , asthma or chronic obstructive pulmonary disease and any disease or condition that in the opinion of the investigator can modify the results of their study is not due to the drug under investigation or that puts the patient at significant risk
* Clinical evidence of immunosuppression (AIDS, hematologic malignancies, use of immunosuppressive drugs and others)
* Patients who received influenza vaccine for the week before inclusion;
* Patients who in the opinion of the attending physician and / or the investigator may need to receive antiviral drugs for treatment of infection with influenza virus A or B (eg, amantadine, rimantadine, oseltamivir, zanamivir)
* Patients who in the opinion of the attending physician and / or the investigator need receive antibacterial drugs for the treatment of acute respiratory infection
* Drug use prior to inclusion by time less than two dose ranges of these drugs (in the case of associations, considered as the reference half-life longer): analgesics, NSAIDs, glucocorticoids and other immunosuppressants, antihistamines, decongestants topical and systemic, as well as any medications that in the opinion of the investigator can modify the results of their study is not due to the drug under investigation or that the interaction place the patient at significant risk
* Having participated in another clinical research for less than a year.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Reduction global symptom score (0-none, 1-weak, 2-medium, 3-strong) | 48 hours
  emergence of adverse events

SECONDARY OUTCOMES:
Use of rescue medication for relief of symptoms, treatment compliance, improvement of foot | 48 hours
  Subjective evaluation of the research subject and the physician

CONTACTS AND LOCATIONS:
Overall Officials: Paulo D Picon, Doctor, Principal Investigator — Federal University of Health Science of Porto Alegre; Luis Felipe C Schmidt, MD, Study Director — Hospital de Clinicas de Porto Alegre; Marisa B Costa, MS, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil